CLINICAL TRIAL: NCT00861887
Title: Comparative Study of 2 Weeks Versus 4 Weeks Treatment With Vancomycin for Clostridium Difficile Colitis
Brief Title: Extended Treatment With Vancomycin for Clostridium Difficile Colitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: Corewell Health East (Other)
Collaborators: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Mihaela Batke, Physician, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIC 2008-173; RC 98690
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2010-01

CONDITIONS: Clostridium Difficile Colitis
Keywords: Clostridium difficile; colitis; recurrence; relapse; Vancomycin
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Colitis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin (Active Comparator): Vancomycin 125 mg every 6 hours x 4 weeks
  Interventions: Drug: Standard Vancomycin; Drug: Extended Vancomycin
- Placebo (Placebo Comparator): Vancomycin 125 mg every 6 hours x 2 weeks, followed by placebo every 6 hours x 2 weeks
  Interventions: Drug: Standard Vancomycin

INTERVENTIONS:
Drug: Standard Vancomycin — Vancomycin treatment 125 mg po every 6 hours x 2 weeks
Drug: Extended Vancomycin — Vancomycin 125 mg every 6 hours x 2 weeks
  Arms: Vancomycin

SUMMARY:
BACKGROUND: Clostridium difficile-associated colitis is an infection of the large bowel, usually associated with previous use of antibiotics. The disease course may be complicated by fulminant disease requiring removal of the colon or by multiple recurrences requiring re-hospitalization. The incidence and severity of Clostridium difficile infection is rising, and it poses an increasing burden on the health system. For example, in one of our previous studies we found that 804 in-patients and 568 out-patients had a positive test for Clostridium difficile toxin at Beaumont Laboratories in 2003. The standard treatment is a 2 week course of Vancomycin or Metronidazole. The clinical response to Metronidazole appears to be declining, and many practicing clinicians prefer Vancomycin as a first-line treatment. The recurrence rate after the treatment is similar for Vancomycin and Metronidazole and is usually in the range of 15-25%, although recent reports noted a recurrence rate up to 50% during outbreaks with a virulent strain. Recently, it has been suggested that a 2 week duration of treatment might not be adequate in clearing the infection.

Our HYPOTHESIS is that a prolongation of Vancomycin treatment from 2 weeks to 4 weeks will lead to a decrease rate of recurrent Clostridium Difficile colitis.

DETAILED DESCRIPTION:
METHODOLOGY: Patients with a first episode of Clostridium difficile colitis will be offered a prolonged course of Vancomycin. It will be disclosed that this is not the standard of care, but that a prolonged course might decrease the relapse rate. After the initial treatment with Vancomycin 125 mg four times daily, the patients will be randomly assigned to receive either 2 weeks of Vancomycin 125 mg four times daily or 2 weeks of placebo. The placebo solution will be prepared by our pharmacy to match the color and taste of the Vancomycin solution. The initial 2 weeks of therapy for both groups will be dispensed at patients' pharmacy. Patients will be called back at the end of 2 weeks and the blinded-phase drugs will be dispensed by our pharmacy staff.

We will ask permission for a follow-up phone call at the end of treatment (1 month) and at a 3-month interval. The patients will be followed longitudinally for a 3-month period. At the end of the follow-up interval, a review of any new medical records of the patient will be made and the patient will be contacted by phone for further details.

ELIGIBILITY:
Inclusion Criteria:

* First episode of Clostridium difficile colitis, defined by a positive toxin assay plus at least one of the following: diarrhea, toxic megacolon or leukocytosis.

Exclusion Criteria:

* previous diagnosis of Clostridium difficile colitis
* concomitant use of oral Metronidazole, Rifampin, Rifaximin, Nitazoxanide, Sacharromyce boulardii or Lactobacillus spp.
* age less than 18 years-old
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
compare the incidence of recurrent Clostridium difficile-associated colitis (CDAD) after a standard 2 week versus a prolonged 4 week course of treatment with Vancomycin | 3 months

SECONDARY OUTCOMES:
assess the response rate to Vancomycin in patients with the first episode of CDAD | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zar FA, Bakkanagari SR, Moorthi KM, Davis MB. A comparison of vancomycin and metronidazole for the treatment of Clostridium difficile-associated diarrhea, stratified by disease severity. Clin Infect Dis. 2007 Aug 1;45(3):302-7. doi: 10.1086/519265. Epub 2007 Jun 19. PMID 17599306
- [Background] Pepin J, Alary ME, Valiquette L, Raiche E, Ruel J, Fulop K, Godin D, Bourassa C. Increasing risk of relapse after treatment of Clostridium difficile colitis in Quebec, Canada. Clin Infect Dis. 2005 Jun 1;40(11):1591-7. doi: 10.1086/430315. Epub 2005 Apr 25. PMID 15889355